CLINICAL TRIAL: NCT06639906
Title: Can the Presence of Intra-Abdominal Adhesion Be Predicted Preoperatively?
Brief Title: Is Preoperative Prediction of Intra-Abdominal Adhesions Possible?
Status: Recruiting | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Other Study IDs: MCBU-Adhesion
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Adhesions Abdominal; Surgery
Keywords: Intraabdominal Adhesion; Decorin; TGF β1; Gynecological Abdominal Surgery; Prediction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — adhesion tissues and patient blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1:: Patients with intra-abdominal adhesions
- Group 2:

SUMMARY:
In this study, it was aimed to evaluate the presence of intra-abdominal adhesion with biochemical markers before the operation, as well as to determine whether there is a relationship between the severity of adhesion and preoperative blood decorin and TGF β1 levels by examining intra-abdominal adhesions histopathologically.This study was conducted on patients who were hospitalized in the department of gynecology and obstetrics of our hospital between 01.09.2023 and 01.09.2024 (1 year) with laparotomy or laparoscopic abdominal surgery planned for gynecological reasons and who had at least 1 previous cesarean section or a history of previous abdominal surgery (laparoscopy or laparotomy). will be made among patients.

The study is voluntary and patients who meet the appropriate criteria will be informed verbally and written consent will be obtained from the patients. Preoperative blood samples will be taken from each patient included in the study. Patients with no adhesions detected in the abdomen during the operation will constitute the control group, and patients with adhesions detected will constitute the study group. The number of patients is planned to be 26 patients in the case group and 28 patients in the control group. Tissue samples removed from detected intra-abdominal adhesions will be taken for histological examination. The tissue samples obtained will be subjected to routine light microscopy tissue monitoring and embedded in paraffin blocks, 5 micron sections will be taken with a microtome and will be examined with a light microscope after being stained with Hematoxylin Eosin. Adhesions detected intra-abdominally are according to the "peritoneal adhesion index" classification; It will be graded in 4 stages: 0: No adhesion, 1: Thin adhesions, blunt dissection, 2: Dense adhesions, sharp dissection, 3: Dense dense and vascularized adhesions, sharp dissection, injury that can be prevented with difficulty. Thanks to the grading of intra-abdominal adhesions, it will be possible to evaluate not only whether the parameters examined are predictive of intra-abdominal adhesions, but also which degree of adhesions they are more effective in predicting. Whether the presence of intra-abdominal adhesion is predictable will be determined by comparing the decorin and TGF β biomarker levels in preoperative blood samples with the decorin and TGF β immunohistochemistry results in the adhesion tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are hospitalized for gynecological reasons with a planned laparotomy or laparoscopic abdominal surgery
* Patients with at least 1 previous cesarean section or history of previous abdominal surgery (laparoscopy or laparotomy)

Exclusion Criteria:

* Patients who do not agree to participate in the study will not be included in the study.
* Pregnant patients will not be included in the study (so that the physiological changes of pregnancy do not affect the results)
* Presence of preoperative clinical or laboratory findings of infection (such as high fever, tachycardia, leukocytosis, high CRP)
* Presence of hematological or coagulation disorders
* History or presence of cancer treatment
* History or presence of connective tissue disease
* Presence of diabetes
* Being under 18 years of age will be considered as exclusion criteria.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Patients with Intraabdominal Adhesions
Study Population: Patients with Intraabdominal Adhesions
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-01-14 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2026-01-14 (Estimated)

PRIMARY OUTCOMES:
1% Patients's intraabdominal adhesion tissues while surgery. Adhesion tissues Staining will be Measured by decorin and TGF β immunohistochemistry. | Baseline
Patient's blood will measured by decorin and TGF β biochemistry technique. | Baseline

SECONDARY OUTCOMES:
Sociodemographic questions were measured by survey technique. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes